CLINICAL TRIAL: NCT05607602
Title: Does the Presence of Uterine Fibroids Cause Changes in the Blood That Increase the Risk of Clots?
Brief Title: Are Uterine Fibroids Pro-thrombotic?
Status: Active, not recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Hemab ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: 301611
Record Dates: First submitted 2022-10-06; First posted 2022-11-07 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Leiomyoma, Uterine; Thrombosis
MeSH Terms: conditions — Leiomyoma; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Women with uterine fibroids, not requiring any medical or surgical treatment.
  Interventions: Other: Comparison of blood samples between the two groups
- 1a: Women with uterine fibroids undergoing myomectomy or hysterectomy for uterine fibroids
- Group 2: Women with no uterine fibroids or uterine pathology on ultrasound scan
  Interventions: Other: Comparison of blood samples between the two groups

INTERVENTIONS:
Other: Comparison of blood samples between the two groups — In this study we will perform global haemostatic assays such as activated partial thromboplastic time (APTT), and prothrombin time (PT). However, these tests provide information about the haemostatic process until the point of initial fibrin formation and ignore the procedure of thrombin generation[18]. In this study we will perform Thrombin Generation studies, Plasma clot Lysis, and RNA sequencing in addition to standard laboratory tests (APTT, PT, FVIII:C, fibrinogen (using Clauss methods), platelet count, liver and renal function tests.
  Groups: 1; Group 2

SUMMARY:
This study will investigate whether the presence of uterine fibroids is independently associated with a laboratory defined pro-thrombotic phenotype. VTE is associated with significant mortality and morbidity. In addition, treating patients with UF and thrombosis represents a particular challenge as fibroids frequently cause menorrhagia, which is exacerbated by anticoagulation. It is therefore important to recognise and detect risk factors and prevent thrombosis wherever possible. If a pro-thrombotic phenotype is detected in patients with UF as their sole risk factor, then this could justify a new approach to the assessment and risk-management of a very large number of patients and could translate into a reduction in both morbidity and mortality for affected patients.

DETAILED DESCRIPTION:
Uterine Fibroids (UF) are benign uterine tumours, also known as leiomyomas. They are estimated to affect up to 80% of women of reproductive age. UF more commonly occur in women of Afro-Caribbean ethnicity. UF may be asymptomatic or associated with a range of symptoms including menorrhagia, dysmenorrhea, sub-fertility, and pressure symptoms.

An association between Venous Thromboembolic disease and UF has been inferred in case reports, series, and one population-based study. The true prevalence and the full scale of the problem is unknown. As UF are so prevalent, in many women, the apparent association reflects the presence of known risk factors for Venous Thromboembolism (VTE) such as thrombophilia, smoking and significant co-morbidities such as cancer. Thrombosis and UF have also been shown to have common risk factors, such as obesity and age. Hormonal therapies, which are often used to treat the symptoms of UF, can also increase the risk of VTE.

However, in a subset of women with VTE and UF, no thrombophilia or acquired risk factors for VTE can be identified. In most of the reported case studies, bulky tumours cause extrinsic compression of pelvic vessels, venous stasis and thus thrombosis. A clinical case review reported by our centre has identified women with thrombosis and UF that do not cause local venous stasis and no additional risk factors for thrombosis. This suggests that there may be additional pathogenic mechanisms underlying the development of thrombosis in individuals with UF. A second centre has also published a case review, similarly identifying an apparent association between UF and thrombosis in the absence of venous stasis.

Clot structure and function is dictated by the conditions present during fibrin generation. Endogenous thrombin production, cellular components and fibrinogen structure are all implicated in altering clot structure and function. There are several plausible mechanisms via which UF may affect thrombin generation, clot formation and structure to generate a pro-thrombotic state. The fibroid tumours may secrete Transforming Growth Factor ß3 (TGF- ß3) and this appears to influence production of thrombomodulin, antithrombin III and plasminogen activator inhibitor 1, all of which can modify the blood's haemostatic capacity and may result in a pro-thrombotic phenotype.

Alternatively, fibroids may mediate an indirect pro-thrombotic effect by inducing iron deficiency anaemia. Iron deficiency anaemia has been associated in numerous case studies and series with thrombotic events, most commonly cerebral venous thrombosis, but also Pulmonary Embolism (PE) and Deep Vein Thrombosis (DVT). Iron deficiency anaemia may also cause a reactive elevation in erythropoietin thrombocytosis, thrombopoietin and FVIII resulting in enhanced thrombin generation. In the proposed study we will exclude participants with moderate and severe anaemia to identify whether any pro-thrombotic phenotype identified is caused by a mechanism other than anaemia.

A pro-thrombotic phenotype can be identified by several laboratory studies that each assess the quality and function of clots formed. In this study we will perform global haemostatic assays such as activated partial thromboplastic time (APTT), and prothrombin time (PT). However, these tests provide information about the haemostatic process until the point of initial fibrin formation and ignore the procedure of thrombin generation. In this study we will perform Thrombin Generation studies, Plasma clot Lysis, and RNA sequencing in addition to standard laboratory tests (APTT, PT, FVIII:C, fibrinogen (using Clauss methods), platelet count, liver and renal function tests.

2 METHODOLOGY Plasma clot lysis and thrombin generation studies will be carried out in platelet poor plasma (PPP). Therefore, the part played by platelets and fibrinogen, it will allow us to freeze and store the samples so that the tests can be done in batch once all the samples have been collected. This allows for testing to be done homogenously under the same conditions.

2.1 Plasma Clot lysis There is evidence that formation of compact clots, with increased resistance to lysis, predisposes to thrombosis. A pro-thrombotic clot phenotype is characterized by small pore size, low clot permeability, and increased resistance to fibrinolysis. The plasma-based clot formation assay allows for a detailed assessment of fibrin formation and breakdown capacity. The principle is that citrated, platelet-poor plasma (PPP) is mixed with an activator of coagulation (recombinant tissue factor or thrombin), as well as phospholipids and calcium to induce fibrin formation. Simultaneously, tPa or another plasminogen activator is added to induce clot lysis. The assay employs a turbidimetric principle, as the fibrin network is first formed and then lysed in the well, turbidity increases and subsequently decreases. Absorbance is registered continuously over a specified time period (e.g., 1.5 h), resulting in the formation of the clot-lysis curve (Figure 1), from which the following parameters can be derived: time to initial fibrin formation (lag phase), maximum absorbance (peak fibrin concentration in well), integral or area under the clot lysis curve (AUC - net fibrin formation), and time from peak to 50% lysis of the clot (50% lysis time).

Pro-thrombotic laboratory phenotypes detected by these assays have been associated with unprovoked VTE, chronic thromboembolic pulmonary hypertension and post thrombotic syndrome. It has been associated with recurrent PE and may be predictive of recurrent DVT.

2.2 Thrombin Generation Thrombin generation is an established tool for assessing the overall function of the blood clotting system. The whole clotting system is engaged in the generation and subsequent inactivation of thrombin and the sum of these actions results in either a haemostatic or a pro-thrombotic event. The method selected for assessing thrombin generation is Calibrated Automated Thrombography (CAT) which involves using a fluorescent substrate containing calcium to trigger thrombin generation, whilst the software continuously monitors and records thrombin concentration in time. Using the specialized software and calibrator, the fluorescent signal can be visualized as a thrombogram. From this, parameters can be calculated such as lag time, time to peak thrombin level, peak thrombin level, and endogenous thrombin potential (ETP).

2.3 RNA sequencing There is evidence in vitro and in vivo that extracellular RNA, released upon vascular injury, promotes thrombosis by augmenting proteases involved in the contact phase of coagulation. This theory was further demonstrated by Kannemeier et al. (2007) who proved that the administration of RNAase delayed thrombus formation and blood vessel occlusion. Extracellular RNA can be directly quantified by a method known as RNA Sequencing. A more robust, reproducible, and easy-to-use technique has been developed by NanoString Technologies, Inc. called "nCounter". Compared to routine RNA Sequencing, nCounter can quantify smaller amounts of starting RNA (1ng vs. 100ng of total RNA). Samples will be analysed in a NanoString Laboratory as nCounter is a proprietary platform.

ELIGIBILITY:
Inclusion Criteria:

Group 1: 35 patients with ultrasound confirmed uterine fibroids. Group 1a: 35 patients with ultrasound confirmed uterine fibroids requiring myomectomy or hysterectomy.

Group 2: 35 control patients with a normal pelvis on ultrasound Able to provide informed consent

Exclusion Criteria:• Personal history of thrombosis

* Pregnant
* Post- partum (within 6 weeks)
* Surgery within 90 days
* Family history of thrombosis (first degree relative)
* Co-morbidities: cancer, liver impairment, renal impairment, uncontrolled hypertension
* Medication: Oral contraception containing oestrogen, hormone replacement therapy with oral oestrogen, antiplatelet therapy, anticoagulation
* Tranexamic Acid within last 48hrs, Zoladex within the last 33 days
* Smoker
* If anaemia (Hb <110 g/L) is demonstrated on the study sample taken

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 18 - 65 years with uterine fibroids confirmed on ultrasound able to provide informed consent
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess for the presence of a laboratory pro-thrombotic phenotype in patients with UF | 1 day (Snapshot in time)

SECONDARY OUTCOMES:
Assess for normalisation of the pro-thrombotic phenotype post-surgery for uterine fibroids | 6 to 12 weeks post operatively
Assess for a correlation between overall uterine size and fibroid volume and markers of a pro-thrombotic phenotype | 1 day (Snapshot in time)

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No